CLINICAL TRIAL: NCT02804464
Title: The DISCOVER Trial (Diagnosis of Infection in Stem Cell Transplant Patients OVER Time)
Acronym: DISCOVER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karius, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 002-CL-01
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Bone Marrow Transplant Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Demonstrate that the Karius Infectious Disease Diagnostic Sequencing Assay performed on plasma can accurately detect the microbiologic etiology in febrile allogeneic stem-cell transplant patients when compared with standard clinical diagnostics

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients who plan on undergoing an allogeneic stem cell transplant and are admitted to UCSF Medical Center.

Exclusion Criteria:

* Inability to provide informed consent and comply with study-related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being evaluated for a stem-cell transplant at the University of California, San Francisco Hospital will be eligible for this study.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-07; Primary Completion 2022-07 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that the Karius Infectious Disease Diagnostic Sequencing Assay performed on plasma can accurately detect the microbiologic etiology in febrile allogeneic stem-cell transplant patients when compared with standard clinical diagnostics. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chin-Hong, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided